CLINICAL TRIAL: NCT01522313
Title: Retrospective Data Analysis of the Impact of Perioperative Kidney Function on Postoperative Outcome
Brief Title: Influence of Perioperative Kidney Function on Postoperative Outcome
Acronym: NEPHRANEST
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Professor of Anesthesiology, Charite University, Berlin, Germany
Other Study IDs: NEPHRANEST
Record Dates: First submitted 2012-01-23; First posted 2012-01-31 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Renal Insufficiency; Acute Kidney Injury
MeSH Terms: conditions — Renal Insufficiency; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Data of patients anesthetized in the years 2006 to 2012 (Hospital stay: January 2006 - June 2012) will be analysed in the study.

SUMMARY:
This study investigates the influence of perioperative changes in serum creatinine on hospital length of stay and mortality.

ELIGIBILITY:
Inclusion Criteria:

* all patients anesthetized between January 2006 - June 2012

Exclusion Criteria:

* end stage renal disease
* pre-anesthesiologic need of renal replacement therapy
* patients undergoing nephrectomy or kidney transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrsospective analysis of electronic charts of all patients that underwent anesthesia between January 2006 - June 2012 in the Department of Anesthesiology at the Charité - University Medicine Berlin, Campus Charité Mitte und Campus Virchow Klinikum.
Sampling Method: Non-Probability Sample
Enrollment: 39369 (Actual)
Dates: Start 2006-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
hospital length of stay | 1 year
  once per case

SECONDARY OUTCOMES:
all cause in-hospital mortality | 1 year
  occurrence during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Claudia D Spies, MD Prof., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - University Medicine Berlin, Berlin, Germany